CLINICAL TRIAL: NCT00895284
Title: Laparoscopic Hysterectomy With and Without Robotic Assistance: a Randomized Prospective Trial
Brief Title: A Trial on Laparoscopic Hysterectomy Versus Robotic Hysterectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Rosanne Kho MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-008892
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Results first posted 2013-06-28 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-05

CONDITIONS: Hysterectomy
Keywords: robotic; laparoscopic surgical procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robot (Experimental): Robotic hysterectomy
  Interventions: Procedure: Robotic hysterectomy
- Standard (Active Comparator): Standard hysterectomy
  Interventions: Procedure: Standard Hysterectomy

INTERVENTIONS:
Procedure: Robotic hysterectomy — Robotic hysterectomy.
  Arms: Robot
Procedure: Standard Hysterectomy — Standard hysterectomy.
  Arms: Standard

SUMMARY:
Robotic technology has been used for laparoscopic hysterectomies for over 10 years. Mayo Clinic Arizona has used robotics in Gynecology for the last 10 years with well over 500 procedures performed. Similar to the laparoscopic approach, small incisions are utilized with the robotic approach. Robotic instruments differ from laparoscopic instruments in that the tips of the instruments can rotate more like the human wrist. The instruments are attached to the robotic arms which are controlled by your surgeon. The surgeon is seated at the surgeon's console which is located 12 feet from the patient while the surgical assistant is at your bedside assisting in the procedure.

This study is being done to compare the procedure times and results after laparoscopic hysterectomies to laparoscopic hysterectomies performed with robotic assistance.

ELIGIBILITY:
Inclusion Criteria:

- All subjects eligible for a laparoscopic hysterectomy with or without bilateral salpingo-oophorectomy, and with or without appendectomy will be recruited.

Exclusion Criteria:

- Patients with malignant disease, pregnancy, gynecologic infection, or requiring procedure on an emergent basis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosanne Kho, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were recruited at Mayo Clinic in Arizona.
Period: Overall Study
Arm/Group | Robot | Standard
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Robot | Standard | Total
Number analyzed (Participants) | 3 | 0 | 3
Age Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 3 |  | 3
  >=65 years | 0 |  | 0
Gender [Number; unit: participants]
  Female | 3 |  | 3
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Total Procedure Time - Skin Incision to Skin Closure
Time Frame: At skin closure.
Population: The study was terminated due to lack of funding; due to the small sample size, no analysis was done.
Arm/Group | Robot | Standard
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Robot | Standard
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated due to lack of funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No